CLINICAL TRIAL: NCT04192266
Title: A Randomized, Double-blind Placebo-controlled Multi-center Study of Identifying Neural Mechanisms of PTSD Symptom Reduction Induced by Combined Estrogen and Prolonged Exposure Therapy
Brief Title: Estrogen and Fear in PTSD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mohammed Milad, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-23-0497; R33MH111907 (NIH); NCT03371654 (obsolete NCT alias)
Record Dates: First submitted 2019-10-17; First posted 2019-12-10 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Estradiol; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prolonged Exposure (PE) therapy with Estradiol (Experimental): A single 2mg dose of estradiol (a form of estrogen) will be taken at home by the study participant 5-6 hours before each of 5 prolonged exposure (PE) therapy treatment sessions (sessions 2 to 6). PE therapy is a validated treatment for PTSD.
  Interventions: Drug: Estradiol; Behavioral: Prolonged Exposure (PE) therapy
- Prolonged Exposure (PE) therapy with Placebo (Placebo Comparator): A single 2mg placebo pill will be taken at home by the study participant 5-6 hours before each of 5 prolonged exposure (PE) therapy treatment sessions (sessions 2 to 6). PE therapy is a validated treatment for PTSD.
  Interventions: Drug: Placebo oral tablet; Behavioral: Prolonged Exposure (PE) therapy

INTERVENTIONS:
Drug: Estradiol — 2.0 mg of estradiol will be taken by mouth by the study participant 5-6 hours before each of 5 PE treatment sessions (Session 2- 6)
  Other Names: Estrace
  Arms: Prolonged Exposure (PE) therapy with Estradiol
Drug: Placebo oral tablet — 2.0 mg placebo pills will be taken by mouth by the study participant 5-6 hours before each of 5 PE treatment sessions ( Sessions 2-6)
  Arms: Prolonged Exposure (PE) therapy with Placebo
Behavioral: Prolonged Exposure (PE) therapy — There will be an introductory Prolonged Exposure (PE) therapy session, followed by 5 imaginal exposure sessions, such that there will be 2 sessions per week conducted for a total of 6 sessions over 3 weeks. The PE sessions are 60 minutes long and consist of imaginal exposure. Specifically, the patient is instructed to imagine the trauma and recount it aloud for about 25-30 minutes. In the following 15 minutes, the patient processes her reactions to revisiting the traumatic event by discussing related thoughts and feelings. The session ends with in vivo exposure homework to be completed that same day as the session. In the last session, imaginal exposure is conducted one last time for the same duration as previous sessions. The therapist and patient review treatment progress and discuss applications of treatment principles to daily life.

SUMMARY:
The purpose of this research study is to determine if taking a pill of estradiol (E2) together with prolonged exposure (PE) therapy can improve this treatment outcome in women diagnosed with Post-Traumatic Stress Disorder (PTSD). 80 subjects will take part in this research study across UTHealth Houston and UPenn (40 subjects at each site). Participants will be randomized into one of two groups, PE + E2 or PE + placebo. The study will include preliminary screening and baseline visits, experimental visits, and therapy visits over the course of six weeks. Several follow-up visits will take place.

DETAILED DESCRIPTION:
Prolonged-exposure (PE) therapy is the treatment of choice for posttraumatic stress disorder (PTSD). Despite its efficacy, a significant number of individuals will not benefit from it or might drop out before the completion of all sessions. This underlies the importance of findings ways to enhance the efficacy of PE in order to improve the life quality of individuals suffering from PTSD. It is now widely accepted that extinction learning paradigms used in fundamental studies are useful laboratory analogs to PE. Studies in healthy controls have suggested that elevated estrogen levels benefit extinction learning by promoting its consolidation and thus enhancing its recall when tested later for it. This is also being reflected by changes in the activation of brain regions forming the fear extinction network, including the amygdala, dorsal anterior cingulate cortex (dACC) and ventromedial prefrontal cortex (vmPFC). It is still unknown whether estradiol (E2) administration can modulate the activation of the fear extinction network in oral contraceptive (OC) users and which E2 dose could yield the best results. During the R61 phase of the study, we found that both doses of E2 were effective in engaging the functional activation of the fear extinction network. Therefore, we will use the lower dose (2mg) for the R33 phase. We will combine E2 administration with PE sessions to see if administration of PE can significantly improve clinical outcomes (reduced PTSD symptoms) and engage the fear extinction network in the brain.

Hypothesis: A general improvement is expected after 3 weeks of treatment in both groups given the anticipated benefits of PE alone. But the benefit of the Estradiol-treated groups is hypothesized be larger; with this group exhibiting significantly higher activation in brain regions associated with fear extinction. This will be noted at the follow-up scan compared to the baseline scan.

PTSD symptom severity expected be significantly lower in the Estradiol and PE group relative to the Placebo+PE group following acute treatment after three weeks of treatment.

The degree of PTSD symptom reduction post- compared to pre-PE after 3 weeks of treatment is expected be associated with BOLD changes in the fear extinction network and reduction in SCR during the extinction recall test after PE. The magnitude of BOLD and SCR changes will be significantly larger in the E2+PE group compared to the Plc+PE group.

ELIGIBILITY:
Inclusion Criteria:

1. Female, 18-45 years of age
2. Chronic (at least one month post-trauma) DSM-5 FULL PTSD diagnosis OR subPTSD diagnosis (subPTSD defined as: meeting criterion A, F, G, H, and clusters B, C, and at least 1 of the clusters D or E.)
3. CAPS-5 Past Month score ≥ 20
4. Criterion A traumatic event
5. Stable medications for 3 or more months by the time of study entrance (with the exception of benzodiazepines)
6. Women on oral contraceptives, specifically those using monophasic or biphasic of first, second, third or fourth generation with up to 35mcg of ethinyl estradiol; OR using etonogestrel / ethinyl estradiol 0.120mg/0.015mg per day vaginal ring birth control; OR using the norelgestromin / ethinyl estradiol 0.150mg/0.035mg per day transdermal patch birth control.
7. Willing and able to provide informed consent

Exclusion Criteria:

1. Diagnosis of bipolar I disorder with a past year manic episode
2. Diagnosis of a psychotic disorder or psychotic symptoms that would interfere with the ability to focus on posttraumatic stress disorder (PTSD) in clinic, as determined by clinical judgment.
3. Diagnosis of moderate or severe substance use disorder that would interfere with the ability to focus on posttraumatic stress disorder (PTSD) in clinic, as determined by clinical judgment.
4. Cognitive impairment that would interfere with the ability to focus on posttraumatic stress disorder (PTSD) in clinic, as determined by clinical judgment.
5. History of neurological disease (that involves the brain), seizure, or significant head trauma (i.e., extended loss of consciousness, neurological sequelae, or known structural brain lesion).
6. Suicidal ideation with imminent risk that warrants a higher level of care.
7. Concurrent trauma focused psychotherapy
8. Pregnancy (to be ruled out by urine ß-HCG).
9. Metallic implants or devices contraindicating magnetic resonance imaging by interfering with patient safety or fMRI data collection. Cases will be cleared by the Principal Investigator and/or Baylor College of Medicine (Imaging).
10. History of breast cancer or hormone-responsive cancer.
11. Use of benzodiazepines
12. Self-injurious behavior that involves suicidal intent, requires medical attention, or occurs daily.
13. High risk of adverse emotional or behavioral reaction, and/or an inability to understand study procedures or the informed consent process, based on investigator/clinician clinical evaluation (e.g., evidence of serious personality disorder, antisocial behavior, serious current stressors, lack of meaningful social support)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Estrogens are female sex hormones that are primarily produced by the ovaries and include estrone (E1), estradiol (E2) and estriol (E3). E2 is the predominant and most potent circulating estrogen produced during the reproductive years in non-pregnant women and is commonly prescribed in pill and transdermal form to treat postmenopausal symptoms
Enrollment: 83 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed R Milad, PhD, Principal Investigator — The University of Texas Health Science Center at Houston (UTHealth Houston); Mohammed R Milad, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania
  - The University of Texas Health Science Center at Houston (UTHealth Houston), Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access and will provide upon reasonable request.
  Requests should be directed to Mohammed.R.Milad@uth.tmc.edu. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 123 participants were screened for eligibility. Of these, 83 participants met inclusion criteria and were enrolled in the study. Among the enrolled participants, 19 withdrew before randomization. The remaining 64 participants were randomized and began study participation.
Period: Overall Study
Arm/Group | Prolonged Exposure (PE) Therapy With Estradiol | Prolonged Exposure (PE) Therapy With Placebo
Started | 31 | 33
Completed | 28 | 31
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prolonged Exposure (PE) Therapy With Estradiol | Prolonged Exposure (PE) Therapy With Placebo | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 33 | 64
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 25 | 29 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 19 | 22 | 41
  More than One Race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 31 | 33 | 64
Marital Status [Count of Participants; unit: Participants]
  Single | 23 | 20 | 43
  Living with Partner | 6 | 7 | 13
  Married | 2 | 3 | 5
  Divorced | 0 | 3 | 3
  Widowed | 0 | 0 | 0
  Separated | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Highest Education Level Completed [Count of Participants; unit: Participants]
  Graduate School | 7 | 11 | 18
  College Graduate | 11 | 13 | 24
  Partial College | 13 | 8 | 21
  High School Graduate | 0 | 1 | 1
  Partial High School | 0 | 0 | 0
  Junior High School | 0 | 0 | 0
  Less than 7 years of school | 0 | 0 | 0
Current Employment Status [Count of Participants; unit: Participants]
  Not applicable | 5 | 1 | 6
  Full-time employment | 11 | 18 | 29
  Part-time employment | 5 | 6 | 11
  Student/Dependent on spouse | 10 | 8 | 18
  Recipient of public/private assistance | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Amygdala Activation as Measured by Functional Magnetic Resonance Imaging (fMRI) Blood Oxygen Level Dependent (BOLD) Signal
Description: Functional Magnetic Resonance Imaging (fMRI) will be used to assess Blood Oxygen Level Dependent (BOLD) signal activation in the amygdala before and after completion of the experimental task. Change in activation will be reported using beta weights; positive beta weights mean greater activation and negative beta weights mean less activation in the specific brain region being monitored
Time Frame: Before and after treatment on Experimental day 2
Population: Data were not collected from 4 participants in the Prolonged Exposure (PE) Therapy With Active Pill arm because 3 participants dropped out and 1 participant had data acquisition errors.
  Data were not collected from 3 participants in the Prolonged Exposure (PE) Therapy With Placebo arm because 2 participants dropped out and 1 participant experienced an adverse event and the visit was not completed.
Measure: Mean (Standard Error); unit: beta weights
Arm/Group | Prolonged Exposure (PE) Therapy With Estradiol | Prolonged Exposure (PE) Therapy With Placebo
Number analyzed (Participants) | 27 | 30
beta weights | 0.534 (0.201) | -0.0037 (0.159)

2. Primary Outcome: Change in Dorsal Anterior Cingulate Cortex (dACC) Activation as Measured by Functional Magnetic Resonance Imaging (fMRI) Blood Oxygen Level Dependent (BOLD) Signal
Description: Functional Magnetic Resonance Imaging (fMRI) will be used to assess Blood Oxygen Level Dependent (BOLD) signal activation in the dorsal anterior cingulate cortex (dACC) before and after completion of the experimental task. Change in activation will be reported using beta weights; positive beta weights mean greater activation and negative beta weights mean less activation in the specific brain region being monitored
Time Frame: Before and after treatment on Experimental day 2
Population: as for outcome 1
Measure: Mean (Standard Error); unit: beta weights
Arm/Group | Prolonged Exposure (PE) Therapy With Estradiol | Prolonged Exposure (PE) Therapy With Placebo
Number analyzed (Participants) | 27 | 30
beta weights | 0.292 (0.213) | -0.0276 (0.219)

3. Primary Outcome: Change in Ventromedial Prefrontal Cortex (vmPFC) Activation as Measured by Functional Magnetic Resonance Imaging (fMRI) Blood Oxygen Level Dependent (BOLD) Signal
Description: Functional Magnetic Resonance Imaging (fMRI) will be used to assess Blood Oxygen Level Dependent (BOLD) signal activation in the ventromedial prefrontal cortex (vmPFC) before and after completion of the experimental task. Change in activation will be reported using beta weights; positive beta weights mean greater activation and negative beta weights mean less activation in the specific brain region being monitored
Time Frame: Before and after treatment on Experimental day 2
Population: as for outcome 1
Measure: Mean (Standard Error); unit: beta weights
Arm/Group | Prolonged Exposure (PE) Therapy With Estradiol | Prolonged Exposure (PE) Therapy With Placebo
Number analyzed (Participants) | 27 | 30
beta weights | 0.512 (0.247) | -0.118 (0.209)

4. Primary Outcome: Change in Hippocampus Activation as Measured by Functional Magnetic Resonance Imaging (fMRI) Blood Oxygen Level Dependent (BOLD) Signal
Description: Functional Magnetic Resonance Imaging (fMRI) will be used to assess Blood Oxygen Level Dependent (BOLD) signal activation in the hippocampus before and after completion of the experimental task. Change in activation will be reported using beta weights; positive beta weights mean greater activation and negative beta weights mean less activation in the specific brain region being monitored.
Time Frame: Before and after treatment on Experimental day 2
Population: as for outcome 1
Measure: Mean (Standard Error); unit: beta weights
Arm/Group | Prolonged Exposure (PE) Therapy With Estradiol | Prolonged Exposure (PE) Therapy With Placebo
Number analyzed (Participants) | 27 | 30
beta weights | 0.341 (0.158) | -0.0606 (0.178)

5. Secondary Outcome: Skin Conductance Response (SCR) During Recall
Description: Skin Conductance Response (SCR) assesses the stress/seat level, or level of anxiety in a particular moment, or in response to a specific cue. SCR are reported in microsiemens, a positive value indicates an increase of response to the condition stimulus relative to 3 seconds prior to its onset. A negative value indicates a decrease in response to the condition stimulus relative to 3 seconds prior to its onset.
Time Frame: Pre - Treatment Experimental Day 2 recall
Population: Data were not collected from 13 participants in the Prolonged Exposure (PE) Therapy With Active Pill arm because 3 participants dropped out, 5 participants had data acquisition errors, and 5 participants had unusable data. Data were not collected from 11 participants in the Prolonged Exposure (PE) Therapy With Placebo arm because 2 dropped out, 2 had data acquisition errors, 1 participant experienced an adverse event and the visit was not completed, and 6 participants had unusable data.
Measure: Mean (Standard Deviation); unit: microsiemens
Arm/Group | Prolonged Exposure (PE) Therapy With Estradiol | Prolonged Exposure (PE) Therapy With Placebo
Number analyzed (Participants) | 18 | 22
microsiemens | -0.0741 (0.0821) | -0.195 (0.0659)

6. Secondary Outcome: Skin Conductance Response (SCR) During Recall
Description: Skin Conductance Response (SCR) assesses the stress/seat level, or level of anxiety in a particular moment, or in response to a specific cue. SCR will be reported in microsiemens
Time Frame: Post- Treatment Experimental Day 2 recall
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: microsiemens
Arm/Group | Prolonged Exposure (PE) Therapy With Estradiol | Prolonged Exposure (PE) Therapy With Placebo
Number analyzed (Participants) | 18 | 22
microsiemens | 0.000479 (0.0167) | 0.0894 (0.0457)

7. Secondary Outcome: Change in PTSD Symptom Assessed by the Clinician-Administered PTSD Scale for DSM-5 (CAPS)
Description: The Clinician-Administered PTSD Scale for DSM-5 (CAPS) measures PTSD symptom severity. CAPS has a total score from 0 to 80, with higher scores indicating more severe PTSD symptoms. The change in score will be reported as the [(Score at 1 month post intervention) - (Score at Baseline)] - A negative value indicates a reduction in PTSD symptom severity
Time Frame: Baseline, 1 month post intervention
Population: Data were not collected from 7 participants in the PE therapy with Estradiol arm: 2 dropped out, 2 are missing baseline and post treatment scores because CAPS was not part of the study at the time and 2 are missing baseline scores because CAPS was not part of the study at this time.
  Data were not collected from 3 participants in the PE therapy with Placebo arm: 2 dropped out and 1 is missing both baseline and post treatment scores because CAPS measure was not part of the study at that time.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Prolonged Exposure (PE) Therapy With Estradiol | Prolonged Exposure (PE) Therapy With Placebo
Number analyzed (Participants) | 24 | 30
score on a scale | -14.83 (1.848) | -18.23 (1.848)

8. Secondary Outcome: Change in PTSD Symptom Assessed by the Clinician-Administered PTSD Scale for DSM-5 (CAPS)
Description: The Clinician-Administered PTSD Scale for DSM-5 (CAPS) measures PTSD symptom severity. CAPS has a total score from 0 to 80, with higher scores indicating more severe PTSD symptoms. The change in score will be reported as the [(Score at 3 month post intervention) - (Score at Baseline)] - A negative value indicates a reduction in PTSD symptom severity
Time Frame: Baseline, 3 months post intervention
Population: Data were not collected from 8 participants in the PE therapy with Estradiol arm: 3 dropped out, 4 are missing baseline scores because CAPS was not part of the study at this time and 1 did not complete the 3 month follow up visit.
  Data were not collected from 3 participants in the PE therapy with Placebo arm: 2 dropped out and 1 is missing baseline scores because CAPS measure was not part of the study at that time.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Prolonged Exposure (PE) Therapy With Estradiol | Prolonged Exposure (PE) Therapy With Placebo
Number analyzed (Participants) | 23 | 30
score on a scale | -21.04 (1.5572) | -22.3 (1.8944)

9. Secondary Outcome: Change in PTSD Symptom Assessed by the Clinician-Administered PTSD Scale for DSM-5 (CAPS)
Description: The Clinician-Administered PTSD Scale for DSM-5 (CAPS) measures PTSD symptom severity. CAPS has a total score from 0 to 80, with higher scores indicating more severe PTSD symptoms. The change in score will be reported as the [(Score at 6 month post intervention) - (Score at Baseline)] - A negative value indicates a reduction in PTSD symptom severity
Time Frame: Baseline, 6 months post intervention
Population: Data were not collected from 8 participants in the PE therapy with Estradiol arm: 3 dropped out, 4 are missing baseline scores because CAPS was not part of the study at this time and 1 did not complete the 6 month follow up visit.
  Data were not collected from 4 participants in the PE therapy with Placebo arm: 2 dropped out and 1 is missing baseline scores because CAPS measure was not part of the study at that time and 1 did not complete the 6 month follow up visit.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Prolonged Exposure (PE) Therapy With Estradiol | Prolonged Exposure (PE) Therapy With Placebo
Number analyzed (Participants) | 23 | 29
score on a scale | -22.83 (1.7812) | -23.62 (1.9095)

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Prolonged Exposure (PE) Therapy With Estradiol | Prolonged Exposure (PE) Therapy With Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33
Other Adverse Events (participants affected / at risk) | 17/31 | 18/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prolonged Exposure (PE) Therapy With Estradiol (N=31) | Prolonged Exposure (PE) Therapy With Placebo (N=33)
nausea and/or vomiting and/or diarrhea (Gastrointestinal disorders) | 4 (4) | 4 (4)
COVID illness or post COVID vaccine symptoms (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (7) — COVID illness or post COVID vaccine symptoms (e.g., ache arm, headache, body ache, prolonged menstruation)
Emotional distress, fatigue (Psychiatric disorders) | 3 (5) | 2 (3)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (4)
Issues related to menstrual cycle (Reproductive system and breast disorders) | 2 (2) | 2 (2) — Issues related to menstrual cycle (e.g., menstrual cramps, spotting, etc.)
Arm bruising and ache (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) — Injury (e.g. work accident, non-suicidal self-injury)
General distress due to Interpersonal Conflict (Social circumstances) | 1 (1) | 1 (1)
Changes in libido (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Weight gain (General disorders) | 0 (0) | 1 (1)
Polyp in uterus found after routine medical checkup (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Concussion (Nervous system disorders) | 0 (0) | 1 (1)
Allergic Reaction (General disorders) | 1 (1) | 0 (0)
Body aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Brain fog and nausea (Nervous system disorders) | 1 (1) | 0 (0)
Fever, nausea, and insomnia (General disorders) | 1 (1) | 0 (0)
Gastrointestinal illness (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lymphangitis (Immune system disorders) | 0 (0) | 1 (1)
Neck pain (General disorders) | 1 (1) | 0 (0)
Tremulousness, headache, nausea (Nervous system disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT04192266/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT04192266/ICF_001.pdf